CLINICAL TRIAL: NCT03789448
Title: MaxART: The Effect of Early Access to ART for All in Swaziland on Economic Outcomes
Brief Title: Early Access to ART for All in Swaziland: Effects on Economic Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Till Bärnighausen (Other)
Collaborators: Clinton Health Access Initiative Inc. (Other)
Responsible Party: Sponsor-Investigator, Till Bärnighausen, University Hospital Heidelberg, University Hospital Heidelberg
Organization: University Hospital Heidelberg (Other)
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: MaxART Economic Evaluation
Record Dates: First submitted 2018-12-16; First posted 2018-12-28 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2019-01

CONDITIONS: HIV/AIDS
Keywords: Antiretroviral Treatment
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Proto-Oncogene Proteins c-raf

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- National HIV Treatment Guidelines (No Intervention): HIV-positive individuals are offered ART per Swaziland's national treatment guidelines
- Early Access to ART for All (Experimental): HIV-positive individuals who are aged 18 years or older are initiated on ART regardless of client's immunological and clinical staging (excluding pregnant or breastfeeding women)
  Interventions: Other: Early Access to ART for All

INTERVENTIONS:
Other: Early Access to ART for All — All HIV-positive individuals will be initiated on Swaziland's recommended first-line ART regimen, unless contraindicated when recommended alternate regimens will be used per national guidelines
  Arms: Early Access to ART for All

SUMMARY:
The purpose of this study is to evaluate the impact of offering early antiretroviral therapy to HIV-positive individuals in government-managed health facilities in Swaziland on a range of economic outcomes

DETAILED DESCRIPTION:
The MaxART study is a three-year stepped-wedge randomized trial with open enrollment for all adults 18 years and older across 14 rural health facilities in Swaziland's Hhohho Region. The main trial registration is accessible at: https://clinicaltrials.gov/ct2/show/record/NCT02909218.

This registration is specific to the economic evaluation of the MaxART study which aims to quantify the causal impacts of early ART initiation (compared to national standard care) on a range of key economic outcomes, including healthcare expenditures, productivity, and household wealth.

ELIGIBILITY:
Inclusion Criteria:

* All HIV-positive individuals who are aged 18 years or older, are ART naïve and attend the health facilities included in the study

Exclusion Criteria:

* All HIV-positive individuals who are <18 years of age
* All HIV-positive pregnant or breastfeeding women
* All HIV-positive individuals who did not consent to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3019 (Actual)
Dates: Start 2014-09-01 (Actual); Primary Completion 2017-08-31 (Actual); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
Total healthcare expenditures (for hospitalization and primary care) | 12 months
  Including direct health care costs (e.g., surgery, medication, consultation) and indirect costs (e.g., transport to clinic, payment for someone to look after children, salary lost for time off...)
Total productivity hours | 24 hours
  Total Hours per day spent on income generation activities

SECONDARY OUTCOMES:
Rate of participants with current employment | At study completion, an average of 1.5 years
  Employment rate among participants, including full-time and part-time salary work
Total sum of self-reported monthly expenditures of the participant's household | 12 months
  Including food and non-food items (e.g., electricity, water, transport, personal care items, insurance, festivals, etc.)
Household Assets Ownership and Living Standards Index | At study completion, an average of 1.5 years
  Aggregated index based on ownership of assets (e.g., refrigerator, TV, table, phone...) and living standards (e.g., flush toilet, cooking facilites, floor/wall/roof material...), total scale score is determined via principal component analysis and averaged around 0

REFERENCES:
- [Derived] Briggs J, Teyssier N, Nankabirwa JI, Rek J, Jagannathan P, Arinaitwe E, Bousema T, Drakeley C, Murray M, Crawford E, Hathaway N, Staedke SG, Smith D, Rosenthal PJ, Kamya M, Dorsey G, Rodriguez-Barraquer I, Greenhouse B. Sex-based differences in clearance of chronic Plasmodium falciparum infection. Elife. 2020 Oct 27;9:e59872. doi: 10.7554/eLife.59872. PMID 33107430
- [Derived] Mobegi FM, Leong LE, Thompson F, Taylor SM, Harriss LR, Choo JM, Taylor SL, Wesselingh SL, McDermott R, Ivey KL, Rogers GB. Intestinal microbiology shapes population health impacts of diet and lifestyle risk exposures in Torres Strait Islander communities. Elife. 2020 Oct 19;9:e58407. doi: 10.7554/eLife.58407. PMID 33074097
- [Derived] Steinert JI, Khan S, Mlambo K, Walsh FJ, Mafara E, Lejeune C, Wong C, Hettema A, Ogbuoji O, Vollmer S, De Neve JW, Mazibuko S, Okello V, Barnighausen T, Geldsetzer P. A stepped-wedge randomised trial on the impact of early ART initiation on HIV-patients' economic outcomes in Eswatini. Elife. 2020 Aug 24;9:e58487. doi: 10.7554/eLife.58487. PMID 32831169
- Available data/document: Study Protocol — https://trialsjournal.biomedcentral.com/articles/10.1186/s13063-017-2128-8

DOCUMENTS (1):
  • Statistical Analysis Plan (2018-12-25): https://cdn.clinicaltrials.gov/large-docs/48/NCT03789448/SAP_000.pdf